CLINICAL TRIAL: NCT06974370
Title: Avoiding Radiation Therapy Due to Intracranial Response to Chemotherapy, Targeted Therapy and/or Immuno-ONcology Therapy for Brain Metastases: Pilot Pragmatic Trial (ACTION-Brain Metastases: Pilot Pragmatic Trial)
Brief Title: Avoiding Radiation Therapy Due to Intracranial Response to Chemotherapy, Targeted Therapy and/or Immuno-ONcology Therapy for Brain Metastases: Pilot Pragmatic Trial
Acronym: ACTION-Brain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Anker, Principal Investigayor, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003613/UVMCC2502
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases, Adult; Brain Metastases From Non-small Cell Lung Cancer (NSCLC)
Keywords: Brain Metastases; Radiation Therapy; NSCLC; Quality of Life; FACT-Br; NANO Scale; Pragmatic Trial
MeSH Terms: conditions — Brain Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic Therapy With Surveillance for Brain Metastases (Experimental): Participants with brain metastases from solid tumors will receive standard-of-care systemic therapy expected to have intracranial activity, such as immunotherapy, targeted therapy, or anti-HER2 agents. A re-evaluation brain MRI will be performed 4-8 weeks after starting therapy. If lesions are stable or responding, patients will continue on systemic therapy with MRI surveillance every 3 months. Radiation therapy may be administered only if progression is observed. All participants are managed according to this pathway, regardless of primary tumor type.
  Interventions: Radiation: Active Surveillance

INTERVENTIONS:
Radiation: Active Surveillance — Following systemic therapy, participants will undergo active surveillance with brain MRI every 3 months. Radiation therapy will only be initiated if disease progression is observed on imaging, at the discretion of the treating physician.

SUMMARY:
This pilot pragmatic trial evaluates the feasibility of avoiding radiation therapy in patients with brain metastases who demonstrate an intracranial response to systemic therapy-including immunotherapy, targeted therapy, and/or chemotherapy. The study will prospectively enroll 45 patients, divided into two cohorts: 30 with non-small cell lung cancer (NSCLC) receiving immunotherapy, and 15 with brain metastases from other solid tumors. Eligible participants must have at least one brain metastasis not planned for radiation or surgery and must be initiating or planning to initiate a systemic therapy regimen expected to penetrate the blood-brain barrier and achieve intracranial activity.

All patients will undergo a re-evaluation brain MRI 4-8 weeks after initiating systemic therapy. If lesions are stable or regressing, patients will continue surveillance without radiation. If progression is noted, standard-of-care radiation may be administered at the discretion of the treating physician. The primary objective is to assess 6-month radiation therapy-free survival (RTFS) in NSCLC patients based on PD-L1 expression status. Secondary endpoints include intracranial progression-free survival, overall survival, radiation necrosis rate, and quality of life. This study seeks to inform future trial design and identify patients who may safely avoid brain radiation.

DETAILED DESCRIPTION:
This pilot pragmatic trial evaluates the feasibility of avoiding radiation therapy in patients with brain metastases who demonstrate an intracranial response to systemic therapy-including immunotherapy, targeted therapy, and/or chemotherapy. The study will prospectively enroll 45 patients, divided into two cohorts: 30 with non-small cell lung cancer (NSCLC) receiving immunotherapy, and 15 with brain metastases from other solid tumors. Eligible participants must have at least one brain metastasis not planned for radiation or surgery and must be initiating or planning to initiate a systemic therapy regimen expected to penetrate the blood-brain barrier and achieve intracranial activity.

All patients will undergo a re-evaluation brain MRI 4-8 weeks after initiating systemic therapy. If lesions are stable or regressing, patients will continue surveillance without radiation. If progression is noted, standard-of-care radiation may be administered at the discretion of the treating physician. The primary objective is to assess 6-month radiation therapy-free survival (RTFS) in NSCLC patients based on PD-L1 expression status. Secondary endpoints include intracranial progression-free survival, overall survival, radiation necrosis rate, and quality of life. This study seeks to inform future trial design and identify patients who may safely avoid brain radiation.

Detailed Description Brain metastases are the most common tumors of the central nervous system. Historically, treatment has included surgical resection followed by whole-brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) to prevent recurrence. While effective at achieving local control, radiation therapy-particularly WBRT-carries a significant risk of cognitive decline and radiation necrosis, especially in patients with longer life expectancies.

Recent advances in systemic therapy-including immune checkpoint inhibitors, tyrosine kinase inhibitors, and other targeted agents-have demonstrated meaningful intracranial activity, especially in NSCLC, the most common source of brain metastases. Despite these advances, little prospective data exists on the safety and efficacy of deferring radiation therapy in patients responding to systemic treatment.

This pilot study aims to assess the feasibility of delaying or omitting brain radiation therapy in patients whose brain metastases respond to systemic therapy. It is a prospective, single-institution study enrolling 45 participants across two cohorts: 30 NSCLC patients receiving immunotherapy and 15 patients with brain metastases from other cancer types. Eligible patients must be initiating systemic therapy with agents expected to cross the blood-brain barrier and have at least one brain metastasis not planned for surgical resection or radiation therapy.

Patients will undergo a re-evaluation MRI 4-8 weeks after starting systemic therapy. If metastases are stable or regressing, radiation will be deferred and the patient will enter a structured surveillance protocol with MRIs every 3 months for up to 2 years. If progression is observed, patients may receive radiation therapy per standard of care.

The primary objective is to determine the variability in 6-month RT-free survival (RTFS) in NSCLC patients with brain metastases based on PD-L1 expression.

Secondary objectives include:

Assessing 6-month RTFS in other histologies

Measuring local and distant intracranial progression-free survival

Evaluating intracranial objective response rate using iRANO criteria

Determining the number of metastases avoiding radiation

Measuring overall survival, disease-specific survival, and radiation necrosis rate

Evaluating quality of life using FACT-Br and neurologic function via the NANO scale

The study is exploratory and descriptive, with outcomes expected to inform the design of future cooperative group trials. It also complements ongoing trials like NRG-BN013 by evaluating outcomes in a population managed initially without radiation.

ELIGIBILITY:
Inclusion Criteria:

Pathologically (histologically or cytologically) proven diagnosis of a solid tumor malignancies within 5 years prior to registration. If the original histologic proof of malignancy is greater than 5 years, then more recent pathologic confirmation (e.g., from a systemic site or brain metastasis) or unequivocal imaging confirmation of extracranial metastatic disease (e.g. CT of the chest/abdomen/pelvis, PET/CT, etc.) is required. These scans are considered standard-of-care (SOC) and will not be ordered for research purposes.

Initiation or planning for initiation of systemic therapy to include one or more of the following categories expected to cause an intracranial response:

* Brain penetrant targeted therapies (e.g. tyrosine kinase inhibitors, multikinase inhibitors, EGFR inhibitor, ALK inhibitor, BRAF/MEK inhibitor)
* Checkpoint inhibitor immunotherapy (e.g. PDL-1 inhibitors, PD1 inhibitors, CTLA-4 inhibitors)
* HER2 antibody-drug conjugate (e.g. TDM1, TDX-D)
* Anti-Hormone therapies for Breast Cancer
* Cytotoxic chemotherapy alone may be started initially, but with plan for immunotherapy or eligible targeted therapy noted above before the re-evaluation MRI head

At least 1 brain metastasis that not planned for radiation therapy or surgery.

All brain metastases not planned for resection much be ≤3 cm, with no minimum size required.

Systemic therapy has started within 4 weeks of MRI brain showing new or progressive disease or plan to start systemic therapy within 4 weeks of MRI brain showing new or progressive disease.

Ability to obtain MRI head scans with contrast. All MRI head scans must have slice thickness ≤1.5 mm.

Age ≥ 18 years

KPS >60

Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

No use of the planned new systemic therapy meeting 2.1.2 criteria to address brain metastases within the last 6 months.

Prior radiotherapy to the active brain metastases (partial or whole brain irradiation, or prophylactic cranial irradiation [PCI])

Patients pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants. Negative urine pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal.

Serious medical comorbidities that in the opinion of the investigator would prevent participation in this study.

Known leptomeningeal disease (LMD)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
6-Month Radiation Therapy-Free Survival (RTFS) by PD-L1 Status in NSCLC Patients with Brain Metastases | 6 months from baseline brain MRI
  To determine variability in 6-month RT-free survival (RTFS) in Non-Small Cell Lung Carcinoma (NSCLC) patients with brain metastases depending on PDL-1 status receiving systemic therapy including immunotherapy

SECONDARY OUTCOMES:
6-month RTFS | 6 months from baseline brain MRI
  To determine 6-month RTFS in patients with brain metastases for histologies other than NSCLC receiving systemic therapy expected to have intracranial activity and NSCLC patients receiving systemic therapy other than immunotherapy expected to have intracranial activity

CONTACTS AND LOCATIONS:
Overall Officials: Randall Holcombe, MD, MBA, Study Director — University of Vermont Cancer Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No